CLINICAL TRIAL: NCT00845780
Title: Withdrawal of Amiodarone Treatment Versus Continuation in Successfully Treated Patients With Persistent Atrial Fibrillation. A Randomized Study.
Brief Title: Withdrawal Versus Continuation of Amiodarone in Successfully Treated Patients With Persistent Atrial Fibrillation
Acronym: WISDOM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Prof Dr I.C. Van Gelder, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T377
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; amiodarone; late recurrence atrial fibrillation; adverse events
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- withdrawal amiodarone (Experimental): withdrawal amiodarone afer at least 6 months of sinus rhythm maintenance on amiodarone therapy
  Interventions: Drug: withdrawal or continuation of amiodarone therapy
- continuation amiodarone (Active Comparator): continuation of amiodarone after 6 months of sinus rhythm maintenance on amiodarone therapy
  Interventions: Drug: withdrawal or continuation of amiodarone therapy

INTERVENTIONS:
Drug: withdrawal or continuation of amiodarone therapy — withdrawal or continuation of amiodarone therapy after at least 6 months sinus rhythm maintenance on amiodarone therapy

SUMMARY:
Amiodarone is considered to be the most effective antiarrhythmic drug in the prevention of persistent atrial fibrillation. It can however cause many adverse events, both cardiac and non-cardiac. Long-term maintenance of sinus rhythm after cardioversion is difficult especially because of high recurrence rates during the first month after cardioversion. Duration of atrial fibrillation, type of underlying disease, left ventricular function, left atrial size and age are associated with maintaining sinus rhythm. Early recurrence of atrial fibrillation may be related to a highly arrhythmogenic period due to recovery from electrical remodelling. Late recurrences may be related to other triggers than recovery from electrical remodelling. In this study the investigators want to investigate the effect of amiodarone withdrawal on the occurrence of late relapses of persistent atrial fibrillation. Furthermore, the investigators want to investigate the effect of amiodarone withdrawal on the occurrence of amiodarone related adverse events as well as adverse events related to atrial fibrillation or underlying heart disease. The investigators also want to investigate which patients characteristics are and potential triggers have a prognostic value in the occurence of late relapses after amiodarone withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* history of persistent atrial fibrillation, necessitating at least one electrical cardioversion
* presence of sinus rhythm during the last 6 months, while on amiodarone treatment without adverse events related to amiodarone
* clinically stable
* age > 18 years
* written informed consent

Exclusion Criteria:

* sinus rhythm maintenance is preferable (because of atrial fibrillation related morbidity or any other reason)
* symptomatic heart failure NYHA III or IV
* unstable angina pectoris
* hemodynamically significant valvular disease
* concomitant treatment with other class I or III antiarrhythmic drug
* PCI,CABG, other cardiac surgery or major non-cardiac surgery within the last three months
* recent myocardial infarction (< 3 months)
* presence of any disease that is likely to shorten life expectancy to < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2000-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
occurrence of late relapse of persistent atrial fibrillation | 2 years

SECONDARY OUTCOMES:
difference in occurrence of adverse events (amiodarone and atrial fibrillation/underlying heart disease related) between both strategies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle C. Van Gelder, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands